CLINICAL TRIAL: NCT03353467
Title: A Prospective Clinical Trial of Endoscopic Nasopharyngectomy for Newly Diagnosed Stage I Nasopharyngeal Carcinoma Patients
Brief Title: Endoscopic Nasopharyngectomy for Newly Diagnosed Stage I Nasopharyngeal Carcinoma Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); First People's Hospital of Foshan (Other); Zhongshan People's Hospital, Guangdong, China (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Prof., Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-FXY-055-NPC
Record Dates: First submitted 2017-11-17; First posted 2017-11-27 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Nasopharyngeal Carcinoma; Endoscopic Surgery; Primary Napharyngeal Carcinama; Stage I Nasopharyngeal Cancer
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Nasopharyngeal Neoplasms | interventions — Endoscopy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group in endoscopic surgery (Experimental): Stage I patients were only treated with endoscopic surgery without additional chemotherapy. Endoscopic nasopharyngectomy included endoscopic resection , with or without posterior pedicle nasal mucoperiosteal flap resurfacing the nasopharyngeal defects.
  Interventions: Procedure: Endoscopic surgery
- Group in IMRT (Active Comparator): Stage I patients were only treated with radical intensity-modulated radiotherapy without additional chemotherapy. IMRT was delivered with a dynamic multileaf intensity-modulating collimator (NOMOS, Sewickley, PA) by a slice-by-slice arc rotation approach.
  Interventions: Radiation: Intensity-modulated radiotherapy

INTERVENTIONS:
Procedure: Endoscopic surgery — Endoscopic nasopharyngectomy included endoscopic resection, with or without posterior pedicle nasal mucoperiosteal flap resurfacing the nasopharyngeal defects.
  Arms: Group in endoscopic surgery
Radiation: Intensity-modulated radiotherapy — All of the patients were received irradiation by IMRT. The target volumes were delineated according to a previously described institutional treatment protocol, which is in accordance with the International Commission on Radiation Units and Measurements reports 50 and 62.
  Arms: Group in IMRT

SUMMARY:
Nasopharyngeal carcinoma (NPC) is most prevalent in eastern Asia, with the highest incidence reported among the Cantonese population from the province of Guangdong. Radiotherapy is the cornerstone of initial treatment due to the radiosensitive behavior of NPC and its deep-seated location. Although radiotherapy has achieved satisfactory results, it can also cause some severe adverse events. Currently, surgery is only applied to the treatment of recurrent NPC (rNPC) patients, mainly dominated by the conventional open surgery. However, the traditional surgery was accompanied by high rate of treatment-induced complications and low rate of block removal, which greatly limited the surgical application to the treatment of primary NPC.

With the continuous improvement in surgical techniques, especially the electronic endoscopic system to be used in the surgical treatment recently, endoscopic nasopharyngectomy can largely overcome these shortcomings of traditional surgery mentioned above.

In addition, the investigators retrospectively analyzed the survival outcomes of 9 patients with NPC (all T1N0M0 according to the UICC / AJCC seventh staging) treated with endoscopic nasopharyngectomy in our hospital, with 5-year rate of overall survival, loco-regional-free survival, distant metastasis-free survival of 100%. Therefore, the investigators considered endoscopic nasopharyngectomy for staged I NPC patients feasible.

This study will focus on the survival outcomes and quality of life of the staged I NPC patients treated with endoscopic nasopharyngectomy.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, biopsy-proven World Health Organization (WHO) types II or III NPC; Stage I disease (American Joint Committee on Cancer 7th edition); Between 18 and 70 years old; Adequate bone marrow, liver and renal function; Satisfactory performance status: a score of 0 or 1 using the Eastern Cooperative Oncology Group System; Patients provided signed informed consent.

Exclusion Criteria:

* Evidence of relapse or distant metastasis; History of prior malignancy or previous treatment for NPC; The presence of uncontrolled life-threatening diseases; The investigator considered the patient unable to complete the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3 years
  The event for overall survival (OS) was death from any cause. The duration was calculated from the date of treatment initiation to the date of death or last follow-up.

SECONDARY OUTCOMES:
distant metastasis-free survival | 3 years
  The event for distant metastasis-free survival (DMFS) was distant metastasis. The duration was calculated from the date of treatment initiation to the date of distant metastasis or the last follow-up.
loco-regional relapse-free survival | 3 years
  The event for loco-regional relapse-free survival (LRRFS) was loco-regional recurrence. The duration was calculated from the date of treatment initiation to the date of loco-regional relapse or last follow-up.
the rates of complications | 1 year
  These complications included mucositis, pharyngitis, xerostomia, nasopharyngeal necrosis

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, MD,Ph.D, Study Director — Sun Yat-sen University
Locations (5):
- China (5):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - The First People's Hospital of Foshan, Guangzhou, Guangdong
  - Zhongshan People's Hospital, Zhongshan, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi